CLINICAL TRIAL: NCT05706558
Title: Retrospective Review of Esophageal Cancer at MSKCC
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1631
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer; Esophagus Cancer
Keywords: Esophageal Cancer; Esophagus Cancer; Memorial Sloan Kettering Cancer Center; 16-1631
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Circumferential resection margin (CRM): Participants will have a diagnosis of esophageal carcinoma and residual tumor >1 mm from the CRM
  Interventions: Procedure: Esophagectomy
- Circumferential resection margin (CRM)-close: Participants will have a diagnosis of esophageal carcinoma and residual tumor >0-1 mm from the CRM
  Interventions: Procedure: Esophagectomy
- Circumferential resection margin (CRM)+: Participants will have a diagnosis of esophageal carcinoma and residual tumor at the surgical CRM
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Esophagectomy

SUMMARY:
Residual tumor at the proximal or distal margin after esophagectomy is a known prognostic factor for poor survival outcomes in patients with esophageal cancer; however, the significance of the circumferential resection margin (CRM) remains controversial. In this study, the investigators sought to evaluate the prognostic significance of the CRM in patients with esophageal cancer undergoing resection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal adenocarcinoma (EAC) or esophageal squamous cell carcinoma (ESCC) undergoing esophagectomy
* Pathologic staged T3 tumors (pT3)

Exclusion Criteria:

* Pathologic staged T0-2 (pT0-2) or T4 tumors (pT4)
* Patients with histologic types other than EAC or ESCC, dysplasia or carcinoma in situ without tumor invasion,
* Patients undergoing salvage esophagectomy
* Evidence of distant metastatic disease
* Patients with a positive proximal or distal margin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing esophagectomy for histologically confirmed esophageal adenocarcinoma (EAC) or esophageal squamous cell carcinoma (ESCC) during the period from 2000 to 2019.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
. Preoperative variables associated with overall survival and progression-free survival (measured from date of surgery) | Up to 2 years
  Preoperative variables associated with overall survival and progression-free survival (measured from date of surgery) and the association between patient characteristics, neoadjuvant therapy, and postoperative morbidity.

SECONDARY OUTCOMES:
Overall survival and progression-free survival (measured from date of surgery) | Up to 2 years
  Postoperative outcomes stratified by the type of esophageal cancer surgery performed.
Postoperative outcomes stratified by the time between neoadjuvant therapy and surgery (i.e., delayed or immediate). | Up to 2 years
Survival outcomes stratified by treatment modality (i.e., definitive chemoradiation therapy or trimodality treatment). | Up to 2 years
Survival outcomes stratified by use of adjuvant therapy (i.e., adjuvant therapy or no adjuvant therapy). | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Molena, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org